CLINICAL TRIAL: NCT05943158
Title: Effect of Myoinositol on Serum Asprosin Levels in Pregnant Women
Brief Title: Myoinositol Effect on Asprosin Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Ali Cenk, Associate Professor, Cyprus International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pregnancy ASP
Record Dates: First submitted 2023-06-20; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Pregnancy Related
Keywords: pregnancy; myoinositol; asprosin
MeSH Terms: conditions — Arachnodactyly | interventions — Inositol; Folic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myoinositol+folic acid group (Experimental): This group is given myoinositol+folic acid (inofolic, ITF company, Italy) (myoinositol 4 gram+folic acid 400 micrograms)
  Interventions: Drug: myoinositol and folic acid
- Only folic acid group (Experimental): This group is given only folic acid once a day (400 micrograms a day)
  Interventions: Drug: folic acid

INTERVENTIONS:
Drug: myoinositol and folic acid — The pregnant women were given myoinositol+folic acid starting from initial examination of pregnancy until 24-28 weeks of gestation (time of oral glucose tolerance test)
  Other Names: inofolic, ITF company
  Arms: Myoinositol+folic acid group
Drug: folic acid — The pregnant women were given only folic acid starting from initial examination of pregnancy until 24-28 weeks of gestation (time of oral glucose tolerance test)
  Other Names: folidoce, ITF company
  Arms: Only folic acid group

SUMMARY:
Asprosin is aa adipokine associated with glucose and insulin metabolism. Insulin and glucose metabolism change during pregnancy and studies examining asprosin levels during pregnancy are increasing rapidly. Considering the beneficial effects of myo-inositol to support the physiological pregnancy, recovering and pre-venting adverse maternal and fetal outcomes, we aimed to evaluate the effects of its supplementation on serum asprosin levels in pregnant women.

DETAILED DESCRIPTION:
Asprosin, which was first mentioned in an article in 2016, is a pluripotent adipokine that is a product of profibrillin and its main source is white adipose tissue. It has been observed that asprosin is associated with glucose metabolism, and its plasma level increases after overnight fasting and decreases after feeding. After the demonstration that asprosin increases glucose secretion from the liver, subsequent studies have determined that its serum levels are increased in type 2 diabetes, human and mouse models with insulin resistance, positively correlates with obesity, and high asprosin levels have been associated with metabolic syndrome.

Pregnancy is known to be a diabetogenic process and insulin resistance is increased during gestation. Also, it is known that there is an increase in the production of adipokines during pregnancy. There are a limited number of studies in pregnancy on asprosin which is known to be produced also from the placenta. Studies examining asprosin in pregnancy in the literature mostly examined the relationship between gestational diabetes (GDM). GDM, which is defined as glucose intolerance with variable severity of hyperglycemia that occurs during pregnancy, is the most common metabolic disorder during pregnancy and its prevalence varies between 5-10% according to the patient population examined and the diagnostic test used. In addition, these patients also have impaired insulin secretion. Recently, it has been shown that asprosin levels are increased in the blood of patients with GDM.

Inositol is a polyol structure molecule belonging to the vitamin B complex, which can be produced in many organs in the body and can also be taken from the outside with food. Myo-inositol (MI) is one of the most important of the 9 inositol stereoisomers, and this molecule has been studied many times in the literature in recent years. In the literature, it is stated that inositol supplementation started in the early weeks of pregnancy prevents GDM onset, especially in women in the risk group for developing GDM like obesity, polycystic ovary syndrome, etc.. MI, which is an intracellular second messenger and has insulin-like effects on glucose metabolism, also reduces insulin resistance.

Based on these data in the literature, it can be thought that altered serum asprosin levels during pregnancy may play a role in the pathogenesis of GDM. In addition, it can be suggested that MI, which have proven effects on glucose metabolism, may have an effect on serum levels of asprosin, which is considered a new insulin resistance marker. In this study, we aimed to examine the effect of the MI on serum asprosin levels of women, which was started in the early stages of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women between 18-40 ages

Exclusion Criteria:

* chronic hypertension,
* pre-pregnancy diabetes or a history of GDM in a previous pregnancy,
* multiple pregnancy,
* history of pregnancy-induced hypertension,
* addiction such as smoking or alcohol,
* thyroid or other endocrine diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Serum asprosin levels | between 5-8 weeks of gestation
  First measurement of serum asprosin level at initial examination
Serum asprosin levels | between 24-28 weeks of gestation which the oral glucose tolerance test is done
  Serum asprosin measurement at the time of oral glucose tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- Near East University Faculty of Medicine, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Background] Romere C, Duerrschmid C, Bournat J, Constable P, Jain M, Xia F, Saha PK, Del Solar M, Zhu B, York B, Sarkar P, Rendon DA, Gaber MW, LeMaire SA, Coselli JS, Milewicz DM, Sutton VR, Butte NF, Moore DD, Chopra AR. Asprosin, a Fasting-Induced Glucogenic Protein Hormone. Cell. 2016 Apr 21;165(3):566-79. doi: 10.1016/j.cell.2016.02.063. Epub 2016 Apr 14. PMID 27087445
- [Background] Zhang L, Chen C, Zhou N, Fu Y, Cheng X. Circulating asprosin concentrations are increased in type 2 diabetes mellitus and independently associated with fasting glucose and triglyceride. Clin Chim Acta. 2019 Feb;489:183-188. doi: 10.1016/j.cca.2017.10.034. Epub 2017 Nov 3. PMID 29104036
- [Background] Wang Y, Qu H, Xiong X, Qiu Y, Liao Y, Chen Y, Zheng Y, Zheng H. Plasma Asprosin Concentrations Are Increased in Individuals with Glucose Dysregulation and Correlated with Insulin Resistance and First-Phase Insulin Secretion. Mediators Inflamm. 2018 Mar 20;2018:9471583. doi: 10.1155/2018/9471583. eCollection 2018. PMID 29743813
- [Background] Hong T, Li JY, Wang YD, Qi XY, Liao ZZ, Bhadel P, Ran L, Yang J, Yan B, Liu JH, Xiao XH. High Serum Asprosin Levels Are Associated with Presence of Metabolic Syndrome. Int J Endocrinol. 2021 Mar 2;2021:6622129. doi: 10.1155/2021/6622129. eCollection 2021. PMID 33747078
- [Background] Metzger BE, Buchanan TA, Coustan DR, de Leiva A, Dunger DB, Hadden DR, Hod M, Kitzmiller JL, Kjos SL, Oats JN, Pettitt DJ, Sacks DA, Zoupas C. Summary and recommendations of the Fifth International Workshop-Conference on Gestational Diabetes Mellitus. Diabetes Care. 2007 Jul;30 Suppl 2:S251-60. doi: 10.2337/dc07-s225. No abstract available. PMID 17596481
- [Background] Kleiblova P, Dostalova I, Bartlova M, Lacinova Z, Ticha I, Krejci V, Springer D, Kleibl Z, Haluzik M. Expression of adipokines and estrogen receptors in adipose tissue and placenta of patients with gestational diabetes mellitus. Mol Cell Endocrinol. 2010 Jan 15;314(1):150-6. doi: 10.1016/j.mce.2009.08.002. Epub 2009 Aug 12. PMID 19682537
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2014 Jan;37 Suppl 1:S81-90. doi: 10.2337/dc14-S081. No abstract available. PMID 24357215
- [Background] Coustan DR, Lowe LP, Metzger BE, Dyer AR; International Association of Diabetes and Pregnancy Study Groups. The Hyperglycemia and Adverse Pregnancy Outcome (HAPO) study: paving the way for new diagnostic criteria for gestational diabetes mellitus. Am J Obstet Gynecol. 2010 Jun;202(6):654.e1-6. doi: 10.1016/j.ajog.2010.04.006. PMID 20510967
- [Background] Mulla WR, Henry TQ, Homko CJ. Gestational diabetes screening after HAPO: has anything changed? Curr Diab Rep. 2010 Jun;10(3):224-8. doi: 10.1007/s11892-010-0109-3. PMID 20425586
- [Background] Hoffmann T, Morcos YAT, Janoschek R, Turnwald EM, Gerken A, Muller A, Sengle G, Dotsch J, Appel S, Hucklenbruch-Rother E. Correlation of metabolic characteristics with maternal, fetal and placental asprosin in human pregnancy. Endocr Connect. 2022 Mar 14;11(3):e220069. doi: 10.1530/EC-22-0069. PMID 35148275
- [Background] Baykus Y, Yavuzkir S, Ustebay S, Ugur K, Deniz R, Aydin S. Asprosin in umbilical cord of newborns and maternal blood of gestational diabetes, preeclampsia, severe preeclampsia, intrauterine growth retardation and macrosemic fetus. Peptides. 2019 Oct;120:170132. doi: 10.1016/j.peptides.2019.170132. Epub 2019 Aug 7. PMID 31400492
- [Background] Croze ML, Soulage CO. Potential role and therapeutic interests of myo-inositol in metabolic diseases. Biochimie. 2013 Oct;95(10):1811-27. doi: 10.1016/j.biochi.2013.05.011. Epub 2013 Jun 10. PMID 23764390
- [Background] Unfer V, Carlomagno G, Dante G, Facchinetti F. Effects of myo-inositol in women with PCOS: a systematic review of randomized controlled trials. Gynecol Endocrinol. 2012 Jul;28(7):509-15. doi: 10.3109/09513590.2011.650660. Epub 2012 Feb 1. PMID 22296306
- [Background] Facchinetti F, Cavalli P, Copp AJ, D'Anna R, Kandaraki E, Greene NDE, Unfer V; Experts Group on Inositol in Basic and Clinical Research. An update on the use of inositols in preventing gestational diabetes mellitus (GDM) and neural tube defects (NTDs). Expert Opin Drug Metab Toxicol. 2020 Dec;16(12):1187-1198. doi: 10.1080/17425255.2020.1828344. Epub 2020 Nov 10. PMID 32966143
- [Background] Motuhifonua SK, Lin L, Alsweiler J, Crawford TJ, Crowther CA. Antenatal dietary supplementation with myo-inositol for preventing gestational diabetes. Cochrane Database Syst Rev. 2023 Feb 15;2(2):CD011507. doi: 10.1002/14651858.CD011507.pub3. PMID 36790138
- [Background] Facchinetti F, Appetecchia M, Aragona C, Bevilacqua A, Bezerra Espinola MS, Bizzarri M, D'Anna R, Dewailly D, Diamanti-Kandarakis E, Hernandez Marin I, Kamenov ZA, Kandaraki E, Lagana AS, Monastra G, Montanino Oliva M, Nestler JE, Orio F, Ozay AC, Papalou O, Pkhaladze L, Porcaro G, Prapas N, Soulage CO, Stringaro A, Wdowiak A, Unfer V. Experts' opinion on inositols in treating polycystic ovary syndrome and non-insulin dependent diabetes mellitus: a further help for human reproduction and beyond. Expert Opin Drug Metab Toxicol. 2020 Mar;16(3):255-274. doi: 10.1080/17425255.2020.1737675. Epub 2020 Mar 19. PMID 32129111
- [Derived] Ozay AC, Ozay OE, Edebal OH, Ozay Y, Montanino Oliva M, Dinicola S, Unfer V. Effect of Myo-Inositol Treatment on Serum Asprosin Levels of Pregnant Women: A Prospective Randomized Controlled Pilot Study. J Pregnancy. 2025 Dec 28;2025:8816154. doi: 10.1155/jp/8816154. eCollection 2025. PMID 41497562